CLINICAL TRIAL: NCT07030244
Title: Treatment Outcomes and Predictive Factors of the Effectiveness and Adherence of Moodpep: an Online Self-help Intervention for College Students With Depressive Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Leiden (Other)
Collaborators: VU University of Amsterdam (Other); Maastricht University (Other); Utrecht University (Other); University of Amsterdam (Other); Rotterdam University of Applied Sciences (Other); Erasmus University Rotterdam (Other); Avans University of applied sciences (Unknown); InHolland University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Sanne van Luenen, Principal investigator, Universiteit Leiden
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Effects of Moodpep
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Internet-based Intervention; Depression; Adherence; Predictors; Students; Effectiveness
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: All students will start with Moodpep: a guided online self-help intervention for college students with depressive symptoms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Moodpep (Experimental): Moodpep is an online self-help intervention to reduce depressive symptoms in college students (Garnefski & Kraaij, 2023). The intervention is based on CBT and consists of four main components in eight modules: behavioral activation, relaxation, changing negative cognitions and goal attainment. Students were advised to work on the intervention for one to two hours each week for about six to eight weeks.
  During the intervention, students received coaching via text messages on the platform. Coaches are trained Master's students in clinical psychology and they provided feedback on the assignments that students completed and motivated students to continue the intervention.
  Interventions: Behavioral: Moodpep

INTERVENTIONS:
Behavioral: Moodpep — See arm description

SUMMARY:
Depressive symptoms are prevalent among college students and often remain untreated. E-health interventions may help overcome treatment barriers by offering accessible and flexible support. This study will evaluate the effects of Moodpep, a guided online intervention for college students with depressive symptoms, and will examine predictors of treatment success and adherence.

ELIGIBILITY:
Eligible for Moodpep were students from the participating universities and universities of applied sciences: VU Amsterdam, Leiden University, Maastricht University, Utrecht University, Erasmus University Rotterdam, University of Amsterdam, InHolland University of Applied Sciences, Avans University of Applied Sciences and Rotterdam University of Applied Sciences.

The following inclusion criteria for Moodpep were used:

1. age 16 or older;
2. informed consent was provided;
3. reading Dutch and/or English fluently;
4. having access to a device with internet (e.g., computer, laptop);
5. providing complete data at baseline; and
6. no severe depressive symptoms (PHQ-9 total score > 20) or risk of suicidal behavior (based on 3 questions).

This last criterion was removed on May 9, 2023. After data collection, for statistical and content-related reasons, PhD students were removed from the analysis, just as students below 18 and above 30 years old, students who indicated their gender was other and students who completed less than 1 module of the intervention. This was done because the focus of the study was on students and not PhD students who are employees in the Netherlands, most students are between 18 and 30 years old, not enough students of another gender participated to include them separately in the analyses, and we were interested in the effects of Moodpep for students who started the intervention.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1050 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms (PHQ-9) | T0 (baseline), T1 (6 weeks post-baseline), T2 (6 months post-baseline)
  Patient Health Questionnaire-9 (PHQ-9; Kroenke et al., 2001). Total scores range from 0 to 27 with higher scores indicating more depressive symptoms.

SECONDARY OUTCOMES:
Adherence | T1 (6 weeks post-baseline)
  Number of modules completed (1-8). For the logistic regression analysis, 2 categories will be made: participants who completed 1 module and participants who completed 2-8 modules.
Predictors | T0 (baseline)
  Age, gender (male, female), nationality (Dutch, international), current psychotropic medication use (yes, no), and current psychotherapy (yes, no).

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - VU Amsterdam, Amsterdam
  - Leiden University, Leiden